CLINICAL TRIAL: NCT01834690
Title: Trends of Immunosuppression Therapy and Their Effectiveness in Patients With Liver Transplantation
Brief Title: Uses of Immunosuppression Therapy in Patients With Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Ning Hsu, Clinical Pharmacist, Chang Gung Memorial Hospital
Other Study IDs: 102-0582C
Record Dates: First submitted 2013-04-11; First posted 2013-04-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Evidence of Liver Transplantation
Keywords: Liver transplantation/epidemiology; Liver transplantation/pharmacology; Health status/drug effects; Agents, immunosuppressive agents

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: None Retained — no biospecimens are to be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- liver transplantation recipients: adult liver transplantation recipients (>=20 years at the date of surgery)

SUMMARY:
Conventionally, the outcome of liver transplantation is usually reported in terms of graft and patient survival, medical and surgical complications, but lack of health-related quality of life (HRQOL) that might be associated with immunosuppression complications (e.g., diabetes, hypertension, dyslipidemia, obesity, metabolic syndrome, cardiovascular disease, renal dysfunction, osteoporosis, and de novo malignancy), disease recurrence, and rejections after transplantation.

DETAILED DESCRIPTION:
Specific aims are proposed to achieve in this study:

1. To compare graft and patient survival rate, incidence of treatment-related adverse effects between different patterns of immunosuppression combination among patients received post-liver transplant care in Kaohsiung Chang Gung Memorial Hospital (KCGMH), Taiwan.
2. To quantify the long-term health impacts of immunosuppressive regimens on quality-adjusted life expectancy (QALE), the loss-of-QALE relating to immunosuppression therapy, and types of transplantation.

ELIGIBILITY:
Aim 1:

Inclusion Criteria:

* age at liver transplantation is at least 20 years

Aim 2:

Inclusion Criteria:

* age at liver transplantation is at least 20 years

Exclusion Criteria:

* deceased patient
* cannot obtain inform consent
* age <20 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects: Patients who had liver transplantation in Kaohsiung Chang Gung Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
incidence of graft and patient mortality, treatment-related complications | 5 years
  Patient will be followed from the date of liver transplantation to the occurence of outcome event for 5 years

SECONDARY OUTCOMES:
health-related quality of life | 5 years
  health-related quality of life will be measured by EQ-5D-5L and 15D

OTHER OUTCOMES:
quality-adjusted life expectancy (QALE), loss-of-QALE | 5 years
  QALE:quality-adjusted weight for each health status (measured by EQ-5D)will be multiplied by the survival time and then summed to calculate the number of QALE.
  Loss-of QALE: the life time expectancy (survival function) for thes study cohort will be compared with Taiwan general population of subjects who are age- and gender-matched with study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ning Hsu, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan